CLINICAL TRIAL: NCT02506283
Title: The Effect of Cryotherapy on Recovery and Performance: A Randomized Controlled Double Blind Trial
Brief Title: The Effect of Thermotherapy on Recovery and Performance
Acronym: Cryotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Collaborators: THIM - die internationale Hochschule für Physiotherapie (Other); Vrije Universiteit Brussel (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr.2015-0113
Record Dates: First submitted 2015-05-27; First posted 2015-07-23 (Estimated); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: cryotherapy; recovery; athletic performance; maximum voluntary contraction; rated perceived exertion; delayed onset muscle soreness; jump performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cooling intervention (Experimental): subjects in this study receive a single pre-exercise (3x MVC) or post-exercise intervention (3x 30 counter movement jumps), consisting of an external cooling application (Zamar Therapy CT clinic) applied to both thighs. Both interventions have a duration of 20 minutes and a temperature of 8°C
  Interventions: Device: Zamar Therapy CT clinic
- thermoneutral intervention (Sham Comparator): subjects in the control group receive a single pre-exercise (3x MVC) or post-exercise (3x 30 counter movement jumps) sham intervention, consisting of a 20 minute external thermoneutral application (Zamar Therapy CT clinic) applied to both thighs. Both sham interventions have a duration of 20 minutes and a temperature of 32°C.
  Interventions: Device: Zamar Therapy CT clinic

INTERVENTIONS:
Device: Zamar Therapy CT clinic — Zamar Therapy is a certified medical product (directive 93/42/EEC and ISO 134 85:2012) (www.zamarmedical.com)

SUMMARY:
This study investigates the effects of cooling on the recovery and performance characteristic in young healthy subjects. The study is divided in two projects:

Project A: investigates the effects of 20 min. post-exercise cooling on vertical jump performance and delayed onset muscle soreness and rated perceived exertion.

Project B: investigates the effects of 20 min. pre-exercise cooling on maximal voluntary contraction of the right M. quadriceps femoris and delayed onset muscle soreness and rated perceived exertion.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of a 20 min. external cooling application (+8°C ) versus a external thermo neutral application (+32°C) up to 72 hours post application.

The study is divided in two projects:

Project A: This study is focusing on the recovery process after a max. jump performance (3x30 counter movement jumps). Directly after the exercise subjects receive a cooling or thermo-neutral application. Recovery characteristics measured by vertical jump performance (objective) and delayed onset muscle soreness and rated perceived exertion (subjective) are measured in function of time up to 72 hours post cooling intervention.

Project B: This study is focusing on the effect of 20 min. cooling or thermo-neutral application on the M. quadriceps femoris performance (MVC). After the thermo-application, the 60% endurance MVC is measured by means of surface EMG (OT Bioelettronica 10-750 Hz) in a ergometer chair 90° degrees knee flexion (Cor 1 Bioelettronica). Muscle conduction velocity, MVC (objective), delayed onset muscle soreness and rated perceived exertion (subjective) are measured in function of time up to 72 hours post thermo-application.

ELIGIBILITY:
Inclusion Criteria:

* only healthy young subjects 18-30 years
* no musculoskeletal surgery in trunk and lower extremities
* injury history in trunk and lower extremity for more than one year
* subjects taking anticonceptive medication are allowed to participate

Exclusion Criteria:

* actual injuries or injuries for less than one year in trunk and /or lower extremities
* injury history in trunk and lower extremity for more than one year with complaints
* anxiety of cooling
* subjects on medication
* pace maker
* cardiovascular disease
* pregnancy
* skeletal problems
* appendectomy for less than two years
* Morbus Raynaud syndrome

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-05; Primary Completion 2018-11 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, PhD, Principal Investigator — University of Applied Sciences and Arts of Southern Switzerland SUPSI
Locations (1):
- University of Applied Sciences and Arts of Southern Switzerland SUPSI, Landquart, Kanton Graubünden, Switzerland

REFERENCES:
- [Background] Bleakley C, McDonough S, Gardner E, Baxter GD, Hopkins JT, Davison GW. Cold-water immersion (cryotherapy) for preventing and treating muscle soreness after exercise. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008262. doi: 10.1002/14651858.CD008262.pub2. PMID 22336838
- [Background] Ross ML, Garvican LA, Jeacocke NA, Laursen PB, Abbiss CR, Martin DT, Burke LM. Novel precooling strategy enhances time trial cycling in the heat. Med Sci Sports Exerc. 2011 Jan;43(1):123-33. doi: 10.1249/MSS.0b013e3181e93210. PMID 20508537
- [Result] Ascensao A, Leite M, Rebelo AN, Magalhaes S, Magalhaes J. Effects of cold water immersion on the recovery of physical performance and muscle damage following a one-off soccer match. J Sports Sci. 2011 Feb;29(3):217-25. doi: 10.1080/02640414.2010.526132. PMID 21170794
- [Result] Banfi G, Lombardi G, Colombini A, Melegati G. Whole-body cryotherapy in athletes. Sports Med. 2010 Jun 1;40(6):509-17. doi: 10.2165/11531940-000000000-00000. PMID 20524715
- [Result] Barnett A. Using recovery modalities between training sessions in elite athletes: does it help? Sports Med. 2006;36(9):781-96. doi: 10.2165/00007256-200636090-00005. PMID 16937953
- [Result] Pointon M, Duffield R, Cannon J, Marino FE. Cold application for neuromuscular recovery following intense lower-body exercise. Eur J Appl Physiol. 2011 Dec;111(12):2977-86. doi: 10.1007/s00421-011-1924-1. Epub 2011 Mar 29. PMID 21445604
- [Result] Wegmann M, Faude O, Poppendieck W, Hecksteden A, Frohlich M, Meyer T. Pre-cooling and sports performance: a meta-analytical review. Sports Med. 2012 Jul 1;42(7):545-64. doi: 10.2165/11630550-000000000-00000. PMID 22642829
- [Result] White GE, Wells GD. Cold-water immersion and other forms of cryotherapy: physiological changes potentially affecting recovery from high-intensity exercise. Extrem Physiol Med. 2013 Sep 1;2(1):26. doi: 10.1186/2046-7648-2-26. PMID 24004719
- See also: Zamar thermotherapy — http://www.zamarmedical.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four participants wanted to take part in this study. Two participants had to be excluded due to current pain symptoms.
Groups:
- Single Cooling Intervention: subjects in this study receive a single post-exercise (3x 30 counter movement jumps) recovery intervention, consisting of a 20 minutes external cooling application (Zamar Therapy CT clinic) of 8°C applied to both thighs.
  Zamar Therapy CT clinic: Zamar Therapy is a certified medical product (directive 93/42/EEC and ISO 134 85:2012) (www.zamarmedical.com)
- Single Thermoneutral Intervention: subjects in the control group receive a single post-exercise (3x 30 counter movement jumps) sham intervention, consisting of a 20 minute external thermoneutral application (Zamar Therapy CT clinic) of 32°C applied to both thighs.
  Zamar Therapy CT clinic: Zamar Therapy is a certified medical product (directive 93/42/EEC and ISO 134 85:2012) (www.zamarmedical.com)
Period: Overall Study
Arm/Group | Single Cooling Intervention | Single Thermoneutral Intervention
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Cooling Intervention | Single Thermoneutral Intervention | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (2.3) | 22.4 (1.8) | 22.6 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Delayed-onset Muscle Soreness (DOMS)
Description: The subjective recovery characteristics "Delayed-onset muscle soreness (DOMS)" was rated on a 0-10 cm visual analog scale. DOMS was assessed in a squat position (90° knee angle, with brief holding of maximum 3 seconds) ranging from zero (no soreness) to ten (severe soreness). Higher values mean mean more DOMS and therefore less recovery.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Cooling Intervention | Single Thermoneutral Intervention
Number analyzed (Participants) | 11 | 11
units on a scale
  Baseline | 0.1 (0.0) | 0.1 (0.1)
  0 hours | 5 (1.9) | 4.1 (3.35)
  24 hours | 5.6 (2.2) | 5.0 (2.6)
  48 hours | 7.7 (2.9) | 6.3 (3.2)
  72 hours | 7.7 (3.75) | 6.3 (5.4)

2. Primary Outcome: Ratings of Perceived Exertion (RPE)
Description: The subjective recovery characteristics " Ratings of perceived exertion (RPE)" was rated on a 6-20 Borg scale (from 6 = "no exertion at all" to 20 = "Maximal exertion") in a standing position. The higher value means more exertion and therefore less recovery.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Cooling Intervention | Single Thermoneutral Intervention
Number analyzed (Participants) | 11 | 11
units on a scale
  Baseline | 8 (2) | 7 (2)
  0 hours | 14 (2) | 14 (2)
  24 hours | 9 (3.5) | 8 (2.5)
  48 hours | 12 (5.5) | 8 (4.5)
  72 hours | 11 (3.5) | 7 (4)

3. Primary Outcome: Vertical Jump Performance (VJP)
Description: Vertical jump performance (VJP) was assessed performing three maximal counter mouvemet jumps (CMJs) with a 30-second pause between the three jumps on the Just Jump system (Probotics Inc, Huntsville, AL, USA). The highest jump was recorded.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: height in centimeter
Arm/Group | Single Cooling Intervention | Single Thermoneutral Intervention
Number analyzed (Participants) | 11 | 11
height in centimeter
  Baseline | 38.51 (6.86) | 40.08 (6.99)
  0 hours | 31.02 (7.16) | 35.06 (8.39)
  24 hours | 34.59 (8.07) | 37.82 (7.76)
  48 hours | 29.81 (12.89) | 33.87 (10.81)
  72 hours | 28.44 (13.77) | 33.65 (11.92)

4. Primary Outcome: Peak Power Output (PPO)
Description: Peak power output (PPO) was assessed performing three maximal counter movement jumps (CMJs) on the Just Jump system (Probotics Inc, Huntsville, AL, USA) with a 30-second pause between the three jumps. PPO (presented in watts) was calculated.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: Watt
Arm/Group | Single Cooling Intervention | Single Thermoneutral Intervention
Number analyzed (Participants) | 11 | 11
Watt
  Baseline | 3,375 (876) | 3,267 (636)
  0 hours | 2,920 (855) | 2,963 (702)
  24 hours | 3,137 (953) | 3,130 (677)
  48 hours | 2,846 (1,105) | 2,890 (844)
  72 hours | 2,763 (1,104) | 2,877 (896)

ADVERSE EVENTS:
Time Frame: From Baseline up to 72 hours
Arm/Group | Single Cooling Intervention | Single Thermoneutral Intervention
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT02506283/Prot_SAP_000.pdf